CLINICAL TRIAL: NCT03664167
Title: Weight Loss as Treatment for Gout in Patients With Concomitant Obesity: Protocol for a Proof-of-concept Randomised, Non-blinded, Parallel-group Trial
Brief Title: Weight Loss for Obese Individuals With Gout
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henning Bliddal (Other)
Collaborators: Oak Foundation (Other); The Danish Rheumatism Association (Other); Cambridge Weight Plan Limited (Industry)
Responsible Party: Sponsor-Investigator, Henning Bliddal, Professor, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 140
Record Dates: First submitted 2018-09-07; First posted 2018-09-10 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Gout, Arthritis, Obesity
Keywords: gout; Obesity; arthritis
MeSH Terms: conditions — Gout; Arthritis; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): intensive weight loss diet, with Cambridge weightplan products, and visits to a dietician.
  Interventions: Dietary Supplement: intensive weight loss diet, with Cambridge weightplan products, and visits to a dietician.
- control (No Intervention): usual care

INTERVENTIONS:
Dietary Supplement: intensive weight loss diet, with Cambridge weightplan products, and visits to a dietician. — intensive weight loss diet, with Cambridge weightplan products, and visits to a dietician.
  Arms: intervention

SUMMARY:
This study evaluates effect of weight loss in a group of obese patients with gouty arthritis. The study is a randomised group trial where half the patients receive intensive weight loss in the form of meal replacement from Cambridge as well as supervision from a clinical dietician and the other half get usual care.

DETAILED DESCRIPTION:
Background Gout is an increasingly common disorder characterised by elevated serum urate (SU) and by acute and chronic arthritis causing severe disability and pain. Long-term management of gout focuses on urate-lowering therapy (ULT), and keeping SU under its solubility threshold. When SU is kept under the threshold for solubility, the frequency of gout flares will decrease and the urate crystals dispositioned in the joints will dissolve. New therapeutic management of gout has in recent years emerged. However, despite the potential for effective treatment, gout management remains suboptimal.

there is some physiological evidence, although sparse, that weight loss in patients with gout reduces both SU and number of gout flares. Despite the scarcity of data regarding the effects of weight loss in gout, international guidelines recommend dietary intervention and weight loss as a core management strategy in patients with concomitant gout and obesity The aim with the current study is to address whether or not there is a difference in success rate in weight reduction, SU levels, and possible side-effects between the 2 approaches in the "short-term", by comparing a weight loss group to an ongoing no-treatment (usual care) group.

recruitment Participants will be recruited from the out-patient clinics at the Parker Institute, Bispebjerg and Frederiksberg Hospital and the Department of Rheumatology, Herlev-Gentofte Hospital, Denmark, through advertisements in newspapers and on the website of the Parker Institute. Additionally, local general practitioners will be informed about the possibility to assign patients to the project. All participants will be pre-screened via telephone using a series of standard questions about eligibility according to criteria of inclusion and exclusion. This study aims at being as pragmatic and inclusive as possible with few exclusion criteria

Interventions All the participants who sign informed consent will be randomly assigned to either 16 (8+8) weeks of low-energy diet (LED; 3.4 MJ/day; i.e., the Intensive Diet [ID] group) OR a corresponding 16-week conventional hypo-energetic, high protein diet (app. 5 MJ/day) defined as a control group (i.e., conventional diet [CD] group).

Intensive Diet (ID) Group: The first phase of the study consists of an 8-week weight reduction programme where the participants initiate an LED diet-only, with 3.4 MJ/day (810 kcal per day) in a supervised dietary programme (products provided by The Cambridge Weight Plan). They will be given nutritional and dietetic instructions by an experienced dietitian in sessions of 1-2 h weekly.

The second phase (ID Group) of the study (week 8-16), will consist of an 8 weeks' fixed energy diet programme using 5 MJ/day (1,200 kcal per day) incorporating two diet products daily. The principles of the diet will be in line with the current guidelines for healthy eating issued by the Danish National Board of Health, i.e. low-fat, low-sugar and high-fibre.

Conventional Diet (CD) Group: The programme will consist of a presentation by the same dietitian as for the ID group, who will provide nutritional advice in a 2 h session at baseline (week 0), and in week 8. At these sessions the dietitian will recommend eating ordinary foods in amounts which will provide the patients with approximately 5 MJ/day (1,200 kcal per day). The follow-up meeting at week 16 will not influence the outcome. Thus, during the 16 week trial, the CD group will attend three sessions altogether with a total of approximately 4h of instruction.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of gouty arthritis per expert opinion and the ACR/EULAR 2015 criteria for gout.
* have had at least one self-reported flare in the last 12 months
* BMI >30kg/m2
* >18 years of age

Exclusion Criteria:

* pregnant
* hisotry or suspicion of drug abuse within the past 5 years
* Active muscle disease, cancer, previous kidney disease, and/or fatty liver
* An estimated creatinine clearance <30 mL/min calculated by the Cockcroft-Gault formula using ideal body weight.
* An investigational therapy within 8 weeks or 5 half-lives (whichever is longer) prior to the screening visit.
* Any other medical or psychological condition which, in the opinion of the investigator and/or medical monitor, might create undue risk to the patient or interfere with the patient's ability to comply with the protocol requirements, or to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Bodyweight | 16 weeks
  change in bodyweight (kg) from baseline to week 16 visit.

SECONDARY OUTCOMES:
Serum urate levels. | 16 weeks
  change in serum urate (mg/dL) from baseline to week 16 visit.
Serum urate levels | 16 weeks
  proportion of participants maintaining serum urate levels <6mg/dL at visit week 8 and week 16
Serum urate levels | 16 weeks
  percentage reduction in serum urate(%) at final visit (week 16)
Flare: the proportion of individuals with any gout flare in the FIRST 8 weeks following randomisation] | 8 weeks
  the proportion of individuals with any gout flare in the FIRST 8 weeks following randomisation
Flare:the proportion of individuals with any gout flare in the LAST 8 weeks following randomisation | 16 weeks
  the proportion of individuals with any gout flare in the LAST 8 weeks following randomisation
Flare:the number of gout flares during the trial period for each patient | 16 weeks
  the number of gout flares during the trial period for each patient
functional status - measured by the "Health Assessment Questionaire" (HAQ). | 16 weeks
  change in functional status (HAQ) from baseline to week 16. HAQ consists of 20 questions on disability. The score ranges from 0-3. 0 being without problems and 3 with severe disability. the total score is an average of all questions.
pain from their gout - measured on a visual analoge scale (VAS) | 16 weeks
  change in pain from their gout (VAS) from baseline to week 16. Ranges from 0-100mm on a VAS. 0mm being no pain, 100mm being the worst possible pain.
patient global - measured on a visual analoge scale (VAS) | 16 weeks
  change in patient global (VAS) from baseline to week 16. Ranges from 0-100mm on a VAS. 0mm being best possible health. 100mm being the worst possible health.
fatigue - measured on a visual analoge scale(VAS) | 16 weeks
  change in fatigue (VAS) from baseline to week 16. Ranges from 0-100mm on a VAS. 0mm being no fatigue. 100mm being worst possible fatigue imagined by the patient.
swollen joint count (SJC) | 16 weeks
  chagne in swollen joint count (SJC) from baseline to week 16
tender joint count (TJC) | 16 weeks
  change in tender joint count (TJC) from baseline to week 16
tophi:change in number of tophi from baseline to week 16 | 16 weeks
  change in number of tophi from baseline to week 16
SF-36 | 16 weeks
  change in 36-Item Short Form Health Survey (SF-36: MCS and PCS apply) from baseline to week 16.
  there is included 8 subscales which combine into two overall domains - a physical combined score (PCS) and a mental combined score (MCS). The scales ranges from 0- 100. where 0 is maximum disability and 100 is no disability.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Erik Kristensen, MD, Principal Investigator — CSO The Parker Institute
Locations (1):
- Department of Rheumatology, the Parker Institute, Frederiksberg and Bispebjerg Hospital, Frederiksberg, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2018-08-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT03664167/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-23): https://cdn.clinicaltrials.gov/large-docs/67/NCT03664167/SAP_001.pdf